CLINICAL TRIAL: NCT03488251
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Multiple Dose Regimens of MT-3724 With Gemcitabine and Oxaliplatin for the Treatment of Subjects With Relapsed or Refractory B Cell Non-Hodgkin's Lymphoma
Brief Title: PK,PD,Safety and Tolerability of Multiple Dose Regimens of MT-3724 With Gemcitabine and Oxaliplatin for the Treatment of Patients With Relapsed/Refractory Diffuse Large B Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT-3724_NHL_002
Record Dates: First submitted 2018-03-12; First posted 2018-04-04 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Non-hodgkin Lymphoma,B Cell; Refractory Diffuse Large B-Cell Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX (Experimental): In original protocol and amendment 2, participants will be administered intravenous (IV) MT-3724 10 micrograms per kilograms (mcg/kg) over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants will also be administered Gemcitabine 1000 milligrams per meter square (mg/m^2) as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants will be administered MT-3724 10 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 10 mcg/kg will be administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin will be administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
  Interventions: Drug: MT-3724; Drug: Gemcitabine; Drug: Oxaliplatin
- Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX (Experimental): In original protocol and amendment 2, participants will be planned to administer IV MT-3724 25 mcg/kg over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants will also be planned to administer Gemcitabine 1000 mg/m^2 as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants will be planned to administer MT-3724 25 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 25 mcg/kg will be planned to administer weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin will be planned to administer on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
  Interventions: Drug: MT-3724; Drug: Gemcitabine; Drug: Oxaliplatin
- Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX (Experimental): In original protocol and amendment 2, participants will be planned to administer IV MT-3724 50 mcg/kg over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants will also be planned to administer Gemcitabine 1000 mg/m^2 as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants will be planned to administer MT-3724 50 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 50 mcg/kg will be planned to administer weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin will be planned to administer on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
  Interventions: Drug: MT-3724; Drug: Gemcitabine; Drug: Oxaliplatin
- Part 2: MT-3724/ GEM/ OX (Experimental): Participants will be planned to administer Maximum tolerated dose (MTD) of MT-3724 in combination with Gemcitabine and Oxaliplatin (GEMOX).
  Interventions: Drug: MT-3724; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: MT-3724 — MT-3724 will be administered.
Drug: Gemcitabine — Gemcitabine will be administered.
Drug: Oxaliplatin — Oxaliplatin will be administered.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MT-3724 in combination with gemcitabine and oxaliplatin (GEMOX) in participants with relapsed or refractory B-Cell NHL.

DETAILED DESCRIPTION:
This is a multi-center, open-label two-part study evaluating the safety and tolerability of MT-3724 in combination with GEMOX in relapsed or refractory B-cell Lymphoma patients.

Part 1: (MT-3724 Dose Escalation) Define the maximum tolerated dose (MTD) of MT-3724 in combination with standard treatment of GEMOX

Part 2: (MTD Expansion Cohort) Confirm the safety and tolerability of the MTD of MT-3724 from Part 1 in the MTD Expansion Cohort, where MT-3724 will be given at the MTD in combination with GEMOX. In addition, the PK, PD, immunogenicity and tumor response at the MTD of MT-3724 in combination with GEMOX will be more thoroughly evaluated in Part 2.

In original protocol and amendment 2, participants will be administered intravenous (IV) MT-3724 over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants will also be administered Gemcitabine 1000 milligrams per meter square (mg/m^2) as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants will be administered MT-3724 on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 will be administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin will be administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).

Continued Treatment with MT-3724 in combination with GEMOX will continue for four cycles of until death, disease progression, unacceptable toxicity, withdrawal of consent or another reason for withdrawal.

After four cycles, the participants who experience clinical benefit can continue MT-3724 treatment with additional cycles of 28 days each (either alone or in combination with GEMOX) if supported by the investigator's assessment of the benefit-risk ratio, after consultation with sponsor and Medical Monitor

ELIGIBILITY:
Inclusion Criteria:

1. Be adequately informed about the study and fully consent to participation as demonstrated by signing the written informed consent form before any screening procedure.
2. Be aged ≥18 years on the date of signing the informed consent form.
3. Have relapsed or refractory B-cell NHL that, in the investigator's opinion, could benefit from MT-3724+GEMOX therapy. At least one histologically documented relapse of NHL, by:

   1. Bone marrow biopsy (FNA is not acceptable) or
   2. Excisional lymph node biopsy or
   3. Core biopsy of any involved organ (FNA not acceptable)
   4. CD20-positive histology must have been confirmed at any time during NHL disease course and documented in the medical history
   5. If no histology is available after any relapse the investigator can consult the medical monitor to discuss if the patient can be included
4. All subtypes of B-cell NHL may be considered for Part 1 (MT-3724 dose escalation). Only histologically documented DLBCL (including mixed histology) may be considered for Part 2 (expansion cohort).
5. Have received all approved therapies for NHL that are applicable for the patient in the opinion of the treating physician.

   1. Patients refractory to treatment are eligible.
   2. Patient who have progressed following CAR T-cell therapy are also eligible.
6. Have measurable disease by Lugano Classification for NHL

   1. >1.5 cm longest diameter (LDi) for lymph nodes
   2. >1 cm LDi for extranodal disease
7. Have ECOG performance score of ≤2.
8. Have adequate bone marrow function, as determined by:

   1. Absolute neutrophil count (ANC) ≥1,000/mm3 and
   2. Platelet count ≥50,000 mm³
9. Have adequate kidney function, assessed by thecreatinine clearance (CLcr) to be ≥ 50 mL/min either measured or estimated using the Cockcroft-Gault formula. .

   a. At the investigator's discretion,calculated estimated CLcr of < 50mL/min may be verified eGFR based on the 24-hour urine collection. Subjects with GFR ≥50 mL/min will be eligible irrespective of the estimated CLcr result.
10. Have adequate hepatic function, as determined by:

    1. Total bilirubin ≤1.5 x ULN, or ≤3 x ULN for subjects with Gilbert's Syndrome and
    2. Aspartate aminotransferase (AST) ≤3 x ULN (or ≤ 5.0 x ULN if liver involvement) and
    3. Alanine aminotransferase (ALT) ≤3 x ULN (or ≤ 5.0 x ULN if liver involvement).
11. Have adequate coagulation, as determined by:

    1. INR or PT ≤1.5 x ULN
    2. aPTT ≤1.5 x ULN
12. Have adequate serum albumin, as determined by:

    a. Albumin ≥ 3.0 g/dL
13. Women of reproductive potential must have a negative pregnancy test during the screening period within 72 hours before the start of treatment. Women not of reproductive potential are female subjects who are postmenopausal or permanently sterilized (e.g., tubal occlusion, hysterectomy,bilateral salpingectomy).
14. Subjects of reproductive potential and their partners must agree to either to abstain continuously from heterosexual intercourse or to use a reliable birth control method between signing the informed consent until 6 months following the last dose of MT-3724 or GEMOX . The investigator or a designated associate should advise the subject how to achieve adequate contraception. The following birth control methods may be considered as adequate

    1. Condoms (male or female) with or without a spermicidal agent;
    2. Diaphragm or cervical cap with spermicide;
    3. Intrauterine device;
    4. Hormone-based contraception: Established use of oral, injected, or implanted hormonal methods of contraception;
    5. True abstinence;
    6. Vasectomy is an acceptable method for a male subject or male partner of a female subject.

Exclusion criteria:

1. History or current evidence of neoplastic disease that is histologically distinct from NHL except cervical carcinoma in situ, superficial noninvasive bladder tumors, curatively treated Stage I-II non-melanoma skin cancer, or any other previous cancer curatively treated >2 years before the start of treatment.
2. Current evidence of new or growing brain or spinal metastases during screening.
3. History of allogeneic hematopoietic stem cell transplant within 180 days before the start of treatment.
4. Current evidence of acute or chronic Graft versus Host Disease.
5. Current evidence of CTCAE Grade >1 toxicity (except for hair loss, and those toxicities
6. Current evidence of incomplete recovery from surgery before the start of treatment, or planned surgery at any time during the study until the EoT Visit, except minor elective interventions deemed acceptable by the investigator.
7. History or current evidence of significant (CTCAE Grade ≥2) infection or wound within 4 weeks before the start of treatment.
8. Patients with uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to start of study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis may not be enrolled.
9. Patients with a known history of drug abuse or any chronic neurologic, psychiatric, endocrine, metabolic, immunologic, hepatic or renal disease (including a history of hemolytic uremic syndrome) that in the opinion of the Investigator would adversely affect study participation.
10. Patients with known active Hepatitis C, HIV or a present history of Hepatitis B
11. Women who are pregnant or breastfeeding
12. History or current evidence of hypersensitivity to any study drugs, or current evidence of hypersensitivity requiring systemic steroid doses ≥20 mg/day Prednisone equivalent
13. Received any amount of anti-CD20 MAb therapy within the following periods before the start of treatment

    1. Rituximab (Rituxan®): 84 days; if a subject had received rituximab within 37 Weeks before the start of treatment, then a serum rituximab level must be negative (<500 ng/mL) at the screening period
    2. Obinutuzumab (Gazyva®): 184 days
    3. Ofatumumab (Arzerra®): 88 days
14. Received therapy for NHL (except anti-CD20 Mab listed above) within 4 weeks before the start of treatment
15. Any investigational drug treatment from 4 weeks or 5 half-lives of the agent before the start of treatment, whichever is longer, until the EoT Visit
16. Received radiotherapy to tumor lesions that would be chosen as target lesions (measurable disease) within 4 weeks before the start of treatment, unless the lesion exhibited objective progression between the radiotherapy and the screening according to the Lugano Classification for NHL.

    a. Palliative radiotherapy to non-target lesions is allowed at the investigator's discretion after consultation with the Medical Monitor and sponsor.
17. Received any vaccines within 28 days of the start of treatment, or likely to require vaccines at any time from the start of treatment until 28 days after the last dose of MT-3724. Injectable flu vaccine (inactivated or recombinant) is permitted at the investigator's discretion
18. Received systemic immune modulators within 2 weeks before the start of treatment including but not limited to systemic corticosteroids >20 mg/day of prednisone equivalent, cyclosporine and tacrolimus. Corticosteroids for pre-medication and NSAIDs are permitted.
19. Received any investigational drug treatment within 4 weeks or within 5 half-lives of the therapeutic agent before the start of treatment, whichever is longer, until EoT Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UC Irvine Health / Chao Family Comprehensive Cancer Center, Orange, California
  - Sarcoma Oncology, Santa Monica, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rush University, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Duke Cancer Center, Durham, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - UT Southwestern Medical Center Clinical Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study [Part 1 (Dose Escalation) and Part 2 (Dose Expansion)], to investigate safety, tolerability, efficacy, Pharmacokinetics, Pharmacodynamics and Immunogenicity of MT-3724 in combination with Gemcitabine and Oxaliplatin (GEMOX) in participants with Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma.
Pre-assignment Details: A total of 8 participants were enrolled in the study. This study was terminated in Part 1 as the potential risks outweighed benefits; hence, Part 1 (Cohorts 2 and 3) and Part 2 were not conducted.
Groups:
- Part 1 Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX: In original protocol and amendment 2, participants were administered intravenous (IV) MT-3724 10 micrograms per kilograms (mcg/kg) over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants were also administered Gemcitabine 1000 milligrams per meter square (mg/m^2) as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants were administered MT-3724 10 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 10 mcg/kg was administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin were administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
- Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX: In original protocol and amendment 2, participants were planned to be administered IV MT-3724 25 mcg/kg over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants were also planned to be administered Gemcitabine 1000 mg/m^2 as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants were planned to be administered MT-3724 25 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 25 mcg/kg was planned to be administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin were planned to be administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
- Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX: In original protocol and amendment 2, participants were planned to be administered IV MT-3724 50 mcg/kg over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants were also planned to be administered Gemcitabine 1000 mg/m^2 as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants were planned to be administered MT-3724 50 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 50 mcg/kg was planned to be administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin were planned to be administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
- Part 2: MT-3724/ GEM/ OX: Participants were planned to be administered Maximum tolerated dose (MTD) of MT-3724 in combination with Gemcitabine and Oxaliplatin (GEMOX).
Period: Part 1:Dose Escalation (Up to 168 Days)
Arm/Group | Part 1 Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Started | 8 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Progressive disease | 4 | 0 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 1 | 0 | 0 | 0
Period: Part 2:Dose Expansion (Up to 168 Days)
Arm/Group | Part 1 Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only data for Part 1: Cohort 1 is presented as study was terminated in Part 1 due to premature closure of the trial driven by an unfavorable risk benefit assessment in the concurrent monotherapy study; hence Part 1 (Cohort 2 and 3) and Part 2 were not initiated.
Groups:
- Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX: In original protocol and amendment 2, participants were administered intravenous (IV) MT-3724 10 mcg/kg over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants were also administered Gemcitabine 1000 milligrams per meter square (mg/m^2) as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants were administered MT-3724 10 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 10 mcg/kg was administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin were administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX | Total
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Only data for Part 1: Cohort 1 is presented as study was terminated in Part 1 due to premature closure of the trial driven by an unfavorable risk benefit assessment in the concurrent monotherapy study; hence Part 1 (Cohort 2 and 3) and Part 2 were not initiated.
  Years | 70.8 (7.42) |  |  |  | 70.8 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only data for Part 1: Cohort 1 is presented as study was terminated in Part 1 due to premature closure of the trial driven by an unfavorable risk benefit assessment in the concurrent monotherapy study; hence Part 1 (Cohort 2 and 3) and Part 2 were not initiated.
  Participants
    Female | 1 |  |  |  | 1
    Male | 7 |  |  |  | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Only data for Part 1: Cohort 1 is presented as study was terminated in Part 1 due to premature closure of the trial driven by an unfavorable risk benefit assessment in the concurrent monotherapy study; hence Part 1 (Cohort 2 and 3) and Part 2 were not initiated.
  Participants
    Black or African American | 1 |  |  |  | 1
    White | 6 |  |  |  | 6
    Unknown | 1 |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and 2: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is any treatment-emergent adverse event (TEAE) that occurred after the start of infusion in cycle 1 of Part 1 and the TEAE is at least possibly related to the study drug, as determined by the sponsor after consultation with the investigator(s).
Time Frame: Up to 168 Days
Population: Safety Population consisted of all participants who received at least 1 dose of any study drug (either MT-3724, or gemcitabine or oxaliplatin). Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Participants | 2 |  |  |

2. Primary Outcome: Part 1 and 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is as any untoward medical occurrence in a participant or clinical investigation in a participant administered a pharmaceutical product(s) and which does not necessarily have to have a causal relationship with this experimental intervention(s). A SAE is any AE that is fatal or life-threatening, permanently disabling (incapacitating or interfering with the ability to resume usual life patterns), results in unplanned in-subject hospitalization or prolongation of an existing hospitalization, results in a congenital abnormality or birth defect, or any other situation that require medical or scientific judgement. Number of participants with common >=0 percent (%) TEAEs and SAEs are presented.
Time Frame: Up to 168 Days
Population: Safety Population. Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX: In original protocol and amendment 2, participants were administered intravenous (IV) MT-3724 10 mcg/kg over 1 hour on Days 1, 3, 5, 8, 10 and 12 in Cycles 1 and 2 (each 28-day cycle) and on Days 1, 8, 15, and 22 in Cycles 3 and 4 (each 28-day cycle). Participants were also administered Gemcitabine 1000 milligrams per meter square (mg/m^2) as 30-minute IV infusion and Oxaliplatin 100 mg/m^2 as 2-hour IV infusion on Days 2 and 16 in Cycles 1, 2, 3 and 4 (each 28-day cycle). Per amendment 2, participants were administered MT-3724 10 mcg/kg on Days 1, 3, 5, 8, 10, 12, 15, 22, 29, and 36 in Cycle 1 (42-day cycle). In Cycles 2, 3 and 4, MT-3724 10 mcg/kg was administered weekly on Days 1, 8, 15, and 22 of each 28-day cycle. Gemcitabine and oxaliplatin were administered on Days 16 and 30 of Cycle 1 and on Days 2 and 16 in Cycles 2, 3 and 4 (42-day cycle for Cycle 1 and 28-day cycle for Cycle 2, Cycle 3 and Cycle 4).
Arm/Group | Part 1 Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Participants
  TEAEs | 8 |  |  |
  SAEs | 4 |  |  |

3. Secondary Outcome: Part 1 and 2: Maximum Concentration (Cmax) Following Administration of MT-3724
Description: Blood samples were planned to be collected at indicated time points for pharmacokinetic (PK) analysis of MT-3724. PK Population consisted of all participants who received at least one dose of MT-3724 and have at least one post-Baseline PK value.
Time Frame: Cycle(C)1:Day1:Predose,10 minutes(min) before end of treatment(EOT),5,30 min,1,2,3,4 hours after EOT,Days5,12:Predose,10 min before EOT,5min,2hours after EOT;C2,C3,C4:Day1:Predose,10min before EOT,5 min after EOT(C1 is 42-days;C2,C3,C4 are 28-days cycles)
Population: PK Population. Data was not calculated for Part 1: Cohort 1 due to high proportion of non-quantifiable values (>30% of values were imputed). Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1 Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Micrograms per milliliter | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30% of values were imputed) |  |  |

4. Secondary Outcome: Part 1 and 2: Area Under the Plasma Concentration Time Curve (AUC) Following Administration of MT-3724
Description: Blood samples were planned to be collected at indicated time points for PK analysis of MT-3724.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Hours*micrograms per milliliter | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated due to high proportion of non-quantifiable values (>30% of values were imputed) |  |  |

5. Secondary Outcome: Part 1 and 2: Time to Maximum Plasma Concentration (Tmax) Following Administration of MT-3724
Description: Blood samples were planned to be collected at indicated time points for PK analysis of MT-3724.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Hours | NA [NA to NA] — Median and Full Range could not be calculated due to high proportion of non-quantifiable values (>30% of values were imputed) |  |  |

6. Secondary Outcome: Part 1 and 2: Number of Participants With Immunophenotyping Data Outside the Reference Range
Description: Blood samples were planned to be collected at indicated time points for analysis of immunophenotyping parameters which included cluster of differentiation (CD)3 (Percentage [%] and absolute), CD4 (% and absolute), CD8 (% and absolute), CD4:CD8 ratio, CD19 (% and absolute), Natural Killer (NK) cells (% and absolute), naïve B cells (% and absolute), non-switched memory B cells (% and absolute), class-switched memory B cells, Immunoglobulin (Ig)M only memory B cells (% and absolute), and total memory B cells (% and absolute).
Time Frame: Up to 168 Days
Population: Safety Population. Data was not calculated for Part 1: Cohort 1 as 100% of data was below limit of quantification at all time points. Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Participants | NA — NA indicates that data could not be calculated as 100% of data was below limit of quantification at all time points |  |  |

7. Secondary Outcome: Part 1 and 2: Number of Participants With Anti-drug Antibody Titer
Description: Blood samples were planned to be collected at indicated time points for analysis of anti-drug antibody titer.
Time Frame: Up to 168 Days
Population: Immunogenicity population: All participants who received at least one dose of MT-3724 and have at least one post-Baseline immunogenicity assessment. Data was not calculated for Part 1: Cohort 1 as 100% of data was below limit of quantification at all time points. Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Participants | NA — NA indicates that data could not be calculated as 100% of data was below limit of quantification at all time points |  |  |

8. Secondary Outcome: Part 1 and 2: Number of Participants With Positive Neutralizing Antibodies
Description: Blood samples were planned to be collected at indicated time points for analysis of positive neutralizing antibodies.
Time Frame: Up to 168 Days
Population: Immunogenicity population. Data was not calculated for Part 1: Cohort 1 as 100% of data was below limit of quantification at all time points. Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 8 | 0 | 0 | 0
Participants | NA — NA indicates that data could not be calculated as 100% of data was below limit of quantification at all time points |  |  |

9. Secondary Outcome: Part 1 and 2: Objective Response Rate
Description: Objective response rate is defined as the participants with a reduction in tumor size (Partial Response [PR] or Complete Response [CR]) using the Lugano Classification for Lymphoma, adjusted according to Lymphoma response to immunomodulatory therapy criteria (LYRIC).
Time Frame: Up to 168 Days
Population: Efficacy Population: All participants who received at least 1 dose of any study drug and have the Baseline tumor assessment as well as at least one post-Baseline tumor assessment. Only those participants with data available at the specified time points were analyzed. Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants | 3 |  |  |

10. Secondary Outcome: Part 1 and 2: Disease Control Rate
Description: Disease Control rate is defined as participants with objective response of CR, PR or stable disease (SD) defined as SD for 3 months or longer from the Baseline scan.
Time Frame: Up to 168 Days
Population: Efficacy Population. Only those participants with data available at the specified time points were analyzed. Data could not be calculated for Part 1: Cohort 1 as no participants had a confirmed CR or PR. Data was not collected for Part 1 (Cohorts 2 and 3) and Part 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants | NA — NA indicates that data could not be calculated as no participants had a confirmed CR or PR |  |  |

11. Secondary Outcome: Part 1 and 2: Duration of Response
Description: Duration of Response is defined as the time from first documented stable disease to the actual date of disease progression or death, for participants who met the criteria of having stable disease for at least 3 months from Baseline. Data was not collected due to early termination of the trial.
Time Frame: Up to 168 Days
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 7 | 0 | 0 | 0
Months | NA [NA to NA] — NA indicates that data could not be calculated as no participants had a confirmed CR or PR |  |  |

12. Secondary Outcome: Part 1 and 2: Progression-free Survival
Description: Progression-Free Survival is defined as the time from the start of treatment with MT-3724 on Cycle 1 Day 1 to the date of disease progression or death from any cause. Data was not collected due to early termination of the trial.
Time Frame: Up to 168 Days
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
Number analyzed (Participants) | 7 | 0 | 0 | 0
Months | NA [NA to NA] — NA indicates that data could not be calculated as no participants had a confirmed CR or PR |  |  |

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious TEAEs and SAEs were collected up to 168 days in Part 1.
Description: Safety Population. Only data for Part 1: Cohort 1 is presented as study was terminated in Part 1 due to premature closure of the trial driven by an unfavorable risk benefit assessment in the concurrent monotherapy study; hence Part 1 (Cohort 2 and 3) and Part 2 were not initiated.
Arm/Group | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX | Part 2: MT-3724/ GEM/ OX
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/8 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX (N=8) | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX (N=0) | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX (N=0) | Part 2: MT-3724/ GEM/ OX (N=0)
Capillary leak syndrome (Vascular disorders) | 2 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Chemotherapy induced neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1: MT-3724 10 mcg/kg/ GEM/ OX (N=8) | Part 1: Cohort 2: MT-3724 25 mcg/kg/ GEM/ OX (N=0) | Part 1: Cohort 3: MT-3724 50 mcg/kg/ GEM/ OX (N=0) | Part 2: MT-3724/ GEM/ OX (N=0)
Nausea (Gastrointestinal disorders) | 7 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 5 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Restless leg syndrome (Nervous system disorders) | 2 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 0 | 0
Oedema peripheral (General disorders) | 4 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Early satiety (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 0 | 0 | 0
Platelet count decreased (Investigations) | 4 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 3 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0
Libido increased (Psychiatric disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-popular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT03488251/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT03488251/SAP_001.pdf